CLINICAL TRIAL: NCT02202824
Title: Measuring Beliefs and Norms About Violence Against Women in Rural Uganda: A Randomized Controlled Trial
Brief Title: Measuring Beliefs and Norms About Violence Against Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other)
Responsible Party: Principal Investigator, Alexander Tsai, Assistant in Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: MH096620-S1
Record Dates: First submitted 2014-07-26; First posted 2014-07-29 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Domestic Violence
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Survey questionnaire version 1 (Experimental): Study participants will receive version 1 of the survey questionnaire
  Interventions: Other: Survey questionnaire
- Survey questionnaire version 2 (Experimental): Study participants will receive version 2 of the survey questionnaire
  Interventions: Other: Survey questionnaire
- Survey questionnaire version 3 (Experimental): Study participants will receive version 3 of the survey questionnaire
  Interventions: Other: Survey questionnaire

INTERVENTIONS:
Other: Survey questionnaire — Each of the scale versions elicits personal attitudes toward intimate partner violence and perceived norms about intimate partner violence, in a different fashion

SUMMARY:
The objective of our study was to determine the extent to which contextual information about the circumstances of intimate partner violence affects participants' responses to questions about their personal attitudes toward intimate partner violence.

DETAILED DESCRIPTION:
In national studies conducted throughout sub-Saharan Africa, survey data indicate that there is widespread acceptance of intimate partner violence by both men and women (Alio et al., 2011, Mann & Takyi, 2009, Rani et al., 2004, Uthman et al., 2009). For women, the proximate context of gender-unequal norms has important public health impacts. Men who report beliefs consistent with gender-unequal norms are more likely to be perpetrators of sexual violence (Shannon et al., 2012). Women are more likely to be victimized when they and their partners report concordant beliefs about the acceptability of intimate partner violence (Alio et al., 2011). And finally, women who live in areas characterized by gender-unequal norms about intimate partner violence are at greater risk for having their reproductive health compromised (Hung et al., 2012, Tsai & Subramanian, 2012). Accurate measurement of norms about intimate partner violence therefore has important implications for understanding the health risk environment for women.

The Demographic and Health Surveys (DHS), which are nationally representative surveys conducted worldwide, have served as an important source of information on norms about intimate partner violence. However, a cross-country analysis of DHS data showed that minor deviations in survey wording may account for substantial cross-country variation in the extent to which women provide survey responses consistent with acceptance of intimate partner violence (Yount et al., 2011). Furthermore, in-depth interviews conducted among Bangladeshi women suggest that affirmative responses to DHS-style questions may better reflect their perceptions of prevailing norms or their individualized assumptions about contextual details rather than true beliefs about their acceptance of intimate partner violence (Schuler & Islam, 2008, Schuler et al., 2011). Taken together, these lines of inquiry suggest important limitations in the accuracy with which the DHS measure women's attitudes towards intimate partner violence.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Emancipated minors aged 16-18 years
* Considers Nyakabare Parish their primary place of residence
* Capable of providing informed consent

Exclusion Criteria:

* Minors younger than 18 years, with the exception of emancipated minors
* Does not consider Nyakabare Parish their primary place of residence
* Unable to communicate with research staff, e.g., due to deafness, mutism, or aphasia
* Persons with psychosis, neurological damage, acute intoxication, or an intelligence quotient less than 70, as determined in the field by non-clinical research staff in consultation with a supervisor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1557 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Personal attitudes toward intimate partner violence (5-item scale) | Baseline
Perceived norms about intimate partner violence (5-item scale) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C Tsai, MD, PhD, Principal Investigator — Massachusetts General Hospital; Bernard Kaukhikire, MBA, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

REFERENCES:
- [Derived] Tsai AC, Kakuhikire B, Perkins JM, Vorechovska D, McDonough AQ, Ogburn EL, Downey JM, Bangsberg DR. Measuring personal beliefs and perceived norms about intimate partner violence: Population-based survey experiment in rural Uganda. PLoS Med. 2017 May 23;14(5):e1002303. doi: 10.1371/journal.pmed.1002303. eCollection 2017 May. PMID 28542176